CLINICAL TRIAL: NCT01100320
Title: A Randomized, Open-Label, Single-Center, Single-Dose, Two-Way Crossover Study in Healthy Subjects to Determine the Fed Bioequivalence of Oxycodone Tamper Resistant (OTR) 40-mg Tablets to OxyContin® 40-mg Tablets
Brief Title: A Study to Determine the Fed Bioequivalence of Reformulated OXY Tablets and Original OxyContin® (OXY) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Medical Monitor, Purdue Pharma L.P.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: OTR1004
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy subjects; Opioid
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reformulated OXY 40 mg (Experimental): Reformulated OXY 40 mg x 1 dose
  Interventions: Drug: Reformulated OXY (oxycodone HCl)
- Original OxyContin® (OXY) 40 mg (Active Comparator): Original OxyContin® (OXY) 40 mg x 1 dose
  Interventions: Drug: Original OxyContin® (OXY) (oxycodone HCl)

INTERVENTIONS:
Drug: Reformulated OXY (oxycodone HCl) — Reformulated OXY 40-mg tablet x 1 dose taken with food
  Arms: Reformulated OXY 40 mg
Drug: Original OxyContin® (OXY) (oxycodone HCl) — Original OxyContin® (OXY) 40-mg tablet x 1 dose taken with food
  Arms: Original OxyContin® (OXY) 40 mg

SUMMARY:
To assess the bioequivalence of reformulated OXY tablets (40 mg) relative to the original OxyContin® (OXY) formulation (40 mg) in the fed state.

DETAILED DESCRIPTION:
Oxycodone hydrochloride (oxycodone) is a semi-synthetic opioid analgesic that is effective in the relief of moderate to severe malignant and non-malignant pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 50, inclusive.
* Body weight ranging from 50 to 100 kg and a BMI ≥18 and ≤34 (kg/m2).
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, and ECG.
* Females of child-bearing potential must be using an adequate and reliable method of contraception.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Any history of or current drug or alcohol abuse for 5 years.
* History of or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of an opioid-containing medication in the past 30 days.
* History of known sensitivity to oxycodone, naltrexone, or related compounds.
* Any history of frequent nausea or emesis regardless of etiology.
* Any history of seizures or head trauma with current sequelae.
* Participation in a clinical drug study during the 30 days preceding the initial dose in this study.
* Any significant illness during the 30 days preceding the initial dose in this study.
* Use of any medication including thyroid hormone replacement therapy (hormonal contraception is allowed), vitamins, herbal, and/or mineral supplements, during the 7 days preceding the initial dose.
* Refusal to abstain from food for 4 hours following administration of the study drugs and to abstain from caffeine or xanthine entirely during each confinement.
* Consumption of alcoholic beverages within forty-eight (48) hours of initial study drug administration (Day 1) or anytime following initial study drug administration.
* History of smoking or use of nicotine products within 45 days of study drug administration or a positive urine cotinine test.
* Blood or blood products donated within 30 days prior to administration of the study drugs or anytime during the study, except as required by this protocol.
* Positive results for urine drug screen or alcohol screen at Check-in of each period, and HBsAg, HBsAb (unless immunized), anti-HCV.
* Positive Naloxone HCl challenge test.
* Presence of Gilbert's Syndrome or any known hepatobiliary abnormalities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit - Austin, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22-Jan-2007 (date first ICF signed) to 30-Mar-2007 (last subject follow-up) at 1 site in the US (Austin, TX)
Pre-assignment Details: 174 subjects screened; 84 screen failures; 2 discontinued prior to dosing; 88 randomized and dosed; 14 terminated early; 74 completed.
Groups:
- Reformulated OXY (Test) First: Reformulated OXY 40-mg tablet (test) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations. Subjects in this sequence received Reformulated OXY (Test) in period 1 and Original OxyContin(OXY)(Reference) in period 2.
- Original OxyContin® (OXY) (Reference) First: Original OxyContin® (OXY) 40-mg tablet (reference) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations. Subjects in this sequence received Original OxyContin® (OXY) (Reference)in period 1 and Reformulated OXY (Test) in period 2.
Period: Period 1
Arm/Group | Reformulated OXY (Test) First | Original OxyContin® (OXY) (Reference) First
Started | 43 | 45
Completed | 38 | 38
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Positive Drug Screen | 1 | 1
Not completed — Adverse Event | 2 | 2
Period: Period 2
Arm/Group | Reformulated OXY (Test) First | Original OxyContin® (OXY) (Reference) First
Started | 38 | 38
Completed | 37 | 37
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Randomized Safety Population: Subjects who were randomized, received study drug, and had at least 1 postdose safety assessment.
Arm/Group | Randomized Safety Population
Number analyzed (Participants) | 88
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72-hour period
Population: Full Analysis Population for PK Metrics. Data from all subjects who were randomized, received study drug, and had at least 1 valid PK metric variable were included in the statistical analysis. Subjects who experienced emesis within 12 hours after dosing were excluded from PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Reformulated OXY (Test): Reformulated OXY 40-mg tablet (test) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
- Original OxyContin® (OXY) (Reference): Original OxyContin® (OXY) 40-mg tablet (reference) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 76 | 80
ng/mL | 62.0 (16.5) | 61.5 (12.3)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — A mixed-model analysis of variance was used to compare (test vs reference) and the 90% confidence intervals were estimated for the ratios (test/reference); ANOVA; Geometric Test/Ref Ratio x 100 = 99.9, 90% CI 2-sided [95.40 to 104.52] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

2. Primary Outcome: AUC0-inf - Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 76 | 80
ng*h/mL | 537 (135) | 579 (115)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 92.6, 90% CI 2-sided [90.11 to 95.09] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

3. Primary Outcome: AUC0-t - Area Under Plasma Concentration-time Curve From Time Zero to Time of Last Non-zero Plasma Concentration
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 76 | 80
ng*h/mL | 535 (134) | 577 (115)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 92.6, 90% CI 2-sided [90.13 to 95.13] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

ADVERSE EVENTS:
Time Frame: Ongoing AEs-followed until resolution/30 days after last dose;AEs reported during 7 days following last dose were recorded & followed until resolution,or up to 30 days after last dose.All SAEs were followed until resolution or event/sequelae stabilized.
Description: AEs were learned of through spontaneous reports, subject interview, or subject diaries.
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Serious Adverse Events (participants affected / at risk) | 1/81 | 0/83
Other Adverse Events (participants affected / at risk) | 35/81 | 22/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reformulated OXY (Test) (N=81) | Original OxyContin® (OXY) (Reference) (N=83)
Substance Abuse (positive for cocaine, amphetamine, and MDMA) (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reformulated OXY (Test) (N=81) | Original OxyContin® (OXY) (Reference) (N=83)
Nausea (Gastrointestinal disorders) | 15 (16) | 12 (12) — Systematic and nonsystematic assessments were used for reporting AEs.
Vomiting (Gastrointestinal disorders) | 7 (9) | 4 (4) — Systematic and nonsystematic assessments were used for reporting AEs.
Dizziness (Nervous system disorders) | 5 (6) | 3 (3) — Systematic and nonsystematic assessments were used for reporting AEs.
Headache (Nervous system disorders) | 8 (8) | 3 (3) — Systematic and nonsystematic assessments were used for reporting AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days